CLINICAL TRIAL: NCT03137966
Title: Effect of Deferoxamine on Wound Healing Rate in Patients With Diabetes Foot Ulcers
Acronym: DEFEHU
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Sergiu Catrina, Associated professor, Karolinska University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 170428-DEFEHU
Record Dates: First submitted 2017-04-30; First posted 2017-05-03 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Diabetic Foot Ulcer
Keywords: Diabetes mellitus, foot ulcer, deferoxamine
MeSH Terms: conditions — Diabetic Foot; Diabetes Mellitus; Foot Ulcer | interventions — Deferoxamine

STUDY DESIGN:
Intervention Model Description: prospective, randomised, double-blind and placebo-controlled study with parallel groups, multiple centre trial.
Who Masked: Participant
Masking Description: The drugs (active or placebo) will be supplied by the supervision of Medigelium AB and will have the same appearance.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Deferoxamine (Active Comparator): Patients will be randomised to treatment with Deferoxamine (n=87). Deferoxamine (0.66mg/ml) will be applied locally as a gel (3 times a week) for a period of maximum three months or until intact skin.
  Interventions: Drug: Deferoxamine
- Placebo (Placebo Comparator): Patients will be randomised to treatment with placebo (n=87). Placebo will be applied locally as a gel (3 times a week) for a period of maximum three months or until intact skin.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Deferoxamine — Deferoxamine (0.66mg/ml) will be applied locally as a gel (3 times a week) for a period of maximum three months or until intact skin.
  Other Names: Desferal
  Arms: Deferoxamine
Drug: Placebo — Placebo will be applied locally as a gel (3 times a week) for a period of maximum three months or until intact skin.
  Arms: Placebo

SUMMARY:
Diabetic foot ulcer (DFU) is one of the most invalidating complication of diabetes and represents a big economic burden for the society. No specific therapy is available for diabetic foot ulcers.The aim of this study is to define a new approach for treatment of chronic diabetic wounds. Our concept is based on the improvement of the cellular reaction to hypoxia. It will address the transcriptional factor HIF-1 (Hypoxia inducible factor-1) which is the cellular sensor for oxygen and which is specifically repressed by hyperglycemia. The study will investigate the effect of local deferoxamine (0.66 mg/ml), the only known HIF-1 inducer, on the wound healing rate in patients with neuropathic diabetic foot ulcers. The primary objective of the study will be the reduction with >50% of the wound area after 12 weeks of treatment.

DETAILED DESCRIPTION:
Diabetes is reaching epidemic proportions and is predicted to affect 300 millions people worldwide in 2025. Chronic complications of diabetes represent the main concern for the modern therapy of diabetes and it has become a priority to further characterize their pathophysiological mechanisms to develop novel rational therapeutic strategies. It is a high need to identify additional mechanisms that contribute to the development of chronic complications of diabetes. Today's strategies aiming to improve blood glucose levels have limited efficiency mainly because they induce hypoglycemia when used in the optimal therapeutically range. It is therefore important to develop additional therapeutic strategies that can compensate the relative inefficient blood glucose control. There are other examples where "out of the box thinking" strategies such as treatment of hypertension have shown to be at least as efficient as glucose control to decrease morbidity and mortality in patients with diabetes.

Diabetic foot ulceration represents a major medical, social and economic problem. The lifetime risk of a person with diabetes for developing a foot ulcer is 25% and it is believed that every 30 seconds a lower limb is lost in the world due to diabetes. The condition is also followed by a high 5 years mortality which has been estimated to be 45% after ulceration and 79% after amputation. The mortality of the patients with DFU is worse than the mortality in patients with many common cancers.

The present clinical management for patients with DFU is limited and in consequence 40% of the ulcers are still not healed after one year of treatment. This limited efficacy of the present therapy is the consequence of the relative poor understanding of the pathophysiology of this complication. Even though prolonged exposure of the tissues to hyperglycemia seems to be the primary causative factor for chronic complications of diabetes it has recently become increasingly evident that hypoxia plays an important role in all diabetes complications and especially in chronic diabetic wounds. A low oxygen concentration is the consequence of either a deficient blood supply due to functional circulatory deficiency, micro- and macro-vascular disease but also by a poor local diffusion of the oxygen due to local oedema.

Adaptive responses of cells to hypoxia are mediated by the hypoxia-inducible factor 1 (HIF) which is a heterodimeric transcription factor composed of two subunits, HIF-1 alfa and HIF-1 alfa both of which are constitutively expressed in mammalian cells. Regulation of HIF-1 activity is critically dependent of the degradation of the HIF-1 alfa subunit in normoxia. The molecular basis of its degradation is O2 dependent hydroxylation of at least one of the two proline residues in the oxygen dependent degradation domain (ODDD) of HIF 1-alfa by specific Fe 2+-, oxoglutarate dependent prolyl 4-hydroxylases (HIF hydroxylases). In this form HIF-1 alfa binds to the von Hippel-Lindau (VHL) tumor suppressor protein that acts as an E3 ubiquitin ligase and targets HIF-1 alfa for proteasomal degradation (recently reviewed).

Under hypoxic conditions HIF-1alfa is stabilized against degradation and binds to HRE (hypoxic responsive elements) and up-regulates a series of genes involved in angiogenesis (such as VEGF, angiopoietin-2, -4), glycolytic energy metabolism, cell proliferation and survival which enable the cells to adapt to reduction in oxygen availability . The same induction and activation of HIF-1 can be achieved by inhibiting the degrading enzymes (HIF hydroxylases) with substances that compete with their cofactors i.e. iron or oxoglutarate. Deferoxamine is such a substance which stabilizes and activates HIF-1 by chelating iron.

HIF-1 alfa plays a pivotal role in wound healing, and its expression in the multistage process of normal wound healing has been well characterized. In essence, HIF-1 alfa is necessary for expression of multiple angiogenic growth factors, cell motility and recruitment of endothelial progenitor cells (EPC).

Previous studies have shown that hyperglycemia impairs HIF-1 alfa stability and function. Low levels of HIF-1 alfa expression were also found in foot ulcer biopsies in patients with diabetes. The hypothesis is that the wound healing defect present in diabetes is due to an inhibition of HIF-1. This concept has been demonstrated by showing that local activation of HIF-1 either by two structurally different HIF-hydroxylases inhibitors (deferoxamine and DMOG) or by direct adenovirus mediated transfer of stabile HIF in wounds is followed by improvement of wound healing in diabetic mice (db/db) despite of chronic hyperglycemia. The local activation of HIF induces several pivotal processes for wound healing such as recruitment of the EPCs, angiogenesis, cell migration. Same improvement of wound healing were registered using other methods to induce HIF in the wounds in different animal models.

This study is planned to investigate the efficacy of the local stimulation of HIF for improving wound healing in patients with DFU. It is proposed to use local applied deferoxamine which is the only HIF inducer that is approved for clinical use and has been already tested and proved to be effective in animal models of impaired diabetes on wound healing rate. The dose proposed was evaluated as the most effective in preliminary experiments performed in db/db mice.

ELIGIBILITY:
Inclusion Criteria:

* Chronic foot ulcer (> 1month) (at or below the ankle) grade 1A, 2A (University of Texas Wound Classification System) with an ulcer area between 150-350 mm2.
* No ulcer should present a moderate or severe infection at baseline. Concomitant treatment with systemic antibiotics at baseline is accepted if all ulcers meet none of the criteria defining moderate or severe infection.
* Toe/brachial index >0.6 and/or Tcp02 >50mmHg or ankle/brachial index >0.65, or the pulses at dorsalis pedis/tibialis posterioris clearly palpable.
* If more than one ulcer is present, the largest ulcers that fulfill inclusion criteria will be included
* Patient should be compliant to one of the accepted off-loading system.
* Patients will be able to provide written informed consent

Exclusion Criteria:

* Acute cardiovascular event (myocardial infarction/unstable angina, stroke) within three months prior to randomisation
* Subjects who have undergone vascular reconstruction or angioplasty less than 3 months prior to randomisation
* Decompensated congestive heart failure or functional class 3-4.
* Childbearing potential
* Impaired hepatic function (2 times upper normal limit of ASAT and ALAT)
* Severe renal failure (GFR calculated after Cockcroft's formula <30 ml/min/1.73 m2)
* Ongoing treatment with immunosuppressive drugs
* HbA1c >12 % (108 mmol/l)(12%)
* Polyglobulia (EVF>0.60 men, EVF> 0.56 women)
* Any concomitant disease or condition that may interfere with the possibility for the patient to comply with or complete the study protocol
* Malignancy other than basal-cell carcinoma and cervical carcinoma in situ, requiring any general, local, surgical or radiation therapy.
* History of alcohol or drug abuse
* Osteomyelitis defined as:

  1. There is a clinical suspicion of osteomyelitis;
  2. Ulcer considered for treatment is located at the site of a past amputation;
  3. History of acute osteomyelitis in the past 90 days or history of recurrent osteomyelitis; or
  4. A positive "probe to bone" test.
* Participant in another ongoing study
* Known hypersensitivity to deferoxamine
* Unwillingness to participate following oral and written information
* Subjects with any other severe acute or chronic medical or psychiatric condition that make the subject inappropriate for the study in the judgment of the investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Estimated)
Dates: Start 2022-12-30 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Healing | 3 months
  number of patients who have intact skin healing

SECONDARY OUTCOMES:
Improvement of ulcer | 3 months
  the number of patients who have ulcer healing improvement of > 50%

CONTACTS AND LOCATIONS:
Overall Officials: Sergiu Catrina, MD/Ass.Prof., Principal Investigator — Karolinska University Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Catrina SB, Okamoto K, Pereira T, Brismar K, Poellinger L. Hyperglycemia regulates hypoxia-inducible factor-1alpha protein stability and function. Diabetes. 2004 Dec;53(12):3226-32. doi: 10.2337/diabetes.53.12.3226. PMID 15561954
- [Background] Catrina SB. Impaired hypoxia-inducible factor (HIF) regulation by hyperglycemia. J Mol Med (Berl). 2014 Oct;92(10):1025-34. doi: 10.1007/s00109-014-1166-x. Epub 2014 Jun 12. PMID 25027070
- [Background] Kerr M, Rayman G, Jeffcoate WJ. Cost of diabetic foot disease to the National Health Service in England. Diabet Med. 2014 Dec;31(12):1498-504. doi: 10.1111/dme.12545. Epub 2014 Aug 1. PMID 24984759
- [Background] UK Prospective Diabetes Study Group. Tight blood pressure control and risk of macrovascular and microvascular complications in type 2 diabetes: UKPDS 38. UK Prospective Diabetes Study Group. BMJ. 1998 Sep 12;317(7160):703-13. PMID 9732337
- [Background] Boulton AJ, Vileikyte L, Ragnarson-Tennvall G, Apelqvist J. The global burden of diabetic foot disease. Lancet. 2005 Nov 12;366(9498):1719-24. doi: 10.1016/S0140-6736(05)67698-2. PMID 16291066
- [Background] Apelqvist J, Larsson J, Agardh CD. Long-term prognosis for diabetic patients with foot ulcers. J Intern Med. 1993 Jun;233(6):485-91. doi: 10.1111/j.1365-2796.1993.tb01003.x. PMID 8501419
- [Background] Jeffcoate WJ, Chipchase SY, Ince P, Game FL. Assessing the outcome of the management of diabetic foot ulcers using ulcer-related and person-related measures. Diabetes Care. 2006 Aug;29(8):1784-7. doi: 10.2337/dc06-0306. PMID 16873780
- [Background] Armstrong DG, Wrobel J, Robbins JM. Guest Editorial: are diabetes-related wounds and amputations worse than cancer? Int Wound J. 2007 Dec;4(4):286-7. doi: 10.1111/j.1742-481X.2007.00392.x. No abstract available. PMID 18154621
- [Background] Prompers L, Schaper N, Apelqvist J, Edmonds M, Jude E, Mauricio D, Uccioli L, Urbancic V, Bakker K, Holstein P, Jirkovska A, Piaggesi A, Ragnarson-Tennvall G, Reike H, Spraul M, Van Acker K, Van Baal J, Van Merode F, Ferreira I, Huijberts M. Prediction of outcome in individuals with diabetic foot ulcers: focus on the differences between individuals with and without peripheral arterial disease. The EURODIALE Study. Diabetologia. 2008 May;51(5):747-55. doi: 10.1007/s00125-008-0940-0. Epub 2008 Feb 23. PMID 18297261
- [Background] Cameron NE, Eaton SE, Cotter MA, Tesfaye S. Vascular factors and metabolic interactions in the pathogenesis of diabetic neuropathy. Diabetologia. 2001 Nov;44(11):1973-88. doi: 10.1007/s001250100001. PMID 11719828
- [Background] Jorneskog G, Brismar K, Fagrell B. Pronounced skin capillary ischemia in the feet of diabetic patients with bad metabolic control. Diabetologia. 1998 Apr;41(4):410-5. doi: 10.1007/s001250050923. PMID 9562344
- [Background] Kaelin WG Jr. The von hippel-lindau tumor suppressor protein: an update. Methods Enzymol. 2007;435:371-83. doi: 10.1016/S0076-6879(07)35019-2. PMID 17998064
- [Background] Kaelin WG Jr. The von Hippel-Lindau tumor suppressor protein and clear cell renal carcinoma. Clin Cancer Res. 2007 Jan 15;13(2 Pt 2):680s-684s. doi: 10.1158/1078-0432.CCR-06-1865. PMID 17255293
- [Background] Semenza GL. Life with oxygen. Science. 2007 Oct 5;318(5847):62-4. doi: 10.1126/science.1147949. PMID 17916722
- [Background] Elson DA, Ryan HE, Snow JW, Johnson R, Arbeit JM. Coordinate up-regulation of hypoxia inducible factor (HIF)-1alpha and HIF-1 target genes during multi-stage epidermal carcinogenesis and wound healing. Cancer Res. 2000 Nov 1;60(21):6189-95. PMID 11085544
- [Background] Fadini GP, Sartore S, Schiavon M, Albiero M, Baesso I, Cabrelle A, Agostini C, Avogaro A. Diabetes impairs progenitor cell mobilisation after hindlimb ischaemia-reperfusion injury in rats. Diabetologia. 2006 Dec;49(12):3075-84. doi: 10.1007/s00125-006-0401-6. Epub 2006 Oct 27. PMID 17072586
- [Background] Gao W, Ferguson G, Connell P, Walshe T, Murphy R, Birney YA, O'Brien C, Cahill PA. High glucose concentrations alter hypoxia-induced control of vascular smooth muscle cell growth via a HIF-1alpha-dependent pathway. J Mol Cell Cardiol. 2007 Mar;42(3):609-19. doi: 10.1016/j.yjmcc.2006.12.006. Epub 2006 Dec 21. PMID 17321542
- [Background] Botusan IR, Sunkari VG, Savu O, Catrina AI, Grunler J, Lindberg S, Pereira T, Yla-Herttuala S, Poellinger L, Brismar K, Catrina SB. Stabilization of HIF-1alpha is critical to improve wound healing in diabetic mice. Proc Natl Acad Sci U S A. 2008 Dec 9;105(49):19426-31. doi: 10.1073/pnas.0805230105. Epub 2008 Dec 4. PMID 19057015
- [Background] Thangarajah H, Yao D, Chang EI, Shi Y, Jazayeri L, Vial IN, Galiano RD, Du XL, Grogan R, Galvez MG, Januszyk M, Brownlee M, Gurtner GC. The molecular basis for impaired hypoxia-induced VEGF expression in diabetic tissues. Proc Natl Acad Sci U S A. 2009 Aug 11;106(32):13505-10. doi: 10.1073/pnas.0906670106. Epub 2009 Jul 28. PMID 19666581
- [Background] Hou Z, Nie C, Si Z, Ma Y. Deferoxamine enhances neovascularization and accelerates wound healing in diabetic rats via the accumulation of hypoxia-inducible factor-1alpha. Diabetes Res Clin Pract. 2013 Jul;101(1):62-71. doi: 10.1016/j.diabres.2013.04.012. Epub 2013 May 28. PMID 23726275
- [Background] White RA, Nolan L, Harley D, Long J, Klein S, Tremper K, Nelson R, Tabrisky J, Shoemaker W. Noninvasive evaluation of peripheral vascular disease using transcutaneous oxygen tension. Am J Surg. 1982 Jul;144(1):68-75. doi: 10.1016/0002-9610(82)90604-3. PMID 7091534